CLINICAL TRIAL: NCT03642561
Title: Liver Cancer Institiute ,Fudan University
Brief Title: Evaluation the Treatment Outcome for RFA in Patients With BCLC Stage B HCC in Comparison With TACE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zheng-Gang Ren, zhongshan hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LC-RFA vs.TACE
Record Dates: First submitted 2018-08-08; First posted 2018-08-22 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: group 1 RFA alone group 2 TACE alone
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RFA group (Experimental): Patients in RFA group will accept RFA treatment
  Interventions: Device: radiotherapy ablation
- TACE group (Active Comparator): Patients in TACE group will accept TACE treatment
  Interventions: Device: transarterial chemoembolization(TACE)

INTERVENTIONS:
Device: radiotherapy ablation — We using Cool Tip system or RITA system to perform RFA
  Arms: RFA group
Device: transarterial chemoembolization(TACE) — TACE treatment is a first line treatment for BCLC stage B HCC
  Arms: TACE group

SUMMARY:
Evaluation the Treatment Outcome for RFA in Patients With BCLC Stage B HCC in Comparison With TACE

DETAILED DESCRIPTION:
The investigators conduct this clinical trial to evaluate the treatment outcome of RFA in HCC patients with tumor smaller than 7cm and tumor number less than five ,in comparison with TACE treatment.The primary outcome is overall survival.The secondary outcome is objective response rate.

ELIGIBILITY:
Inclusion criteria:

* age 18 to 75 years ;
* HCC confirmed by pathological or clinical diagnosis according to the American Association for the Study of Liver Diseases criteria ;
* solitary HCC less than 7cm in diameter or multiple HCC lesions less 5
* the absence of portal/hepatic vein invasion, lymph node involvement and extrahepatic metastases;
* lesions visible on ultrasound with a safe path between the lesion and skin;
* an Eastern Cooperative Oncology Group performance status of 0-1;
* Child-Pugh class A or B cirrhosis.

The exclusion criteria :

* received any other previous treatment for HCC;
* severe coagulation disorders;
* evidence of hepatic decompensation including hepatic encephalopathy, ascites as well as esophageal or gastric variceal bleeding;
* presence of serious medical comorbidities, including serious dysfunction of the heart or kidney ;
* currently had other malignancies in addition to HCC.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 60 months

SECONDARY OUTCOMES:
objective response rate | up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhenggang Ren, doctor, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
No plan to make IPDavailable to other researchers